CLINICAL TRIAL: NCT03660813
Title: The Effect of Triggering on the Quantitative Assessment of Follicle Size on Oocyte Development
Brief Title: Follicle Size and Oocyte Development
Acronym: AMJH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4689-17-SMC
Record Dates: First submitted 2018-07-04; First posted 2018-09-07 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: IVF Treatment
Keywords: oocyte, double triggering, follicle size
MeSH Terms: interventions — Chorionic Gonadotropin; Thyrotropin Alfa; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCG triggering (Experimental): Ovitrelle ( hCG 250 mcg)
  Interventions: Diagnostic Test: Follicle measurment; Drug: Ovitrelle ( Hcg 250 mcg)
- Dual triggering (Experimental): Ovitrelle ( Hcg 250 mcg) + Decapeptyl ( GnRH Agonist 0.1 mg*2 )
  Interventions: Diagnostic Test: Follicle measurment; Drug: Ovitrelle ( Hcg 250 mcg); Drug: Decapeptyl ( GnRH Agonist 0.1 mg*2 )

INTERVENTIONS:
Diagnostic Test: Follicle measurment — Follicle will be measured before aspiration
Drug: Ovitrelle ( Hcg 250 mcg) — Drug used for triggering
Drug: Decapeptyl ( GnRH Agonist 0.1 mg*2 ) — Drug used for triggering
  Arms: Dual triggering

SUMMARY:
Studies have shown that the follicles greater in diameter was most likely to have a mature oocyte that was capable of fertilization and best suited for development into a high-quality embryo. Smaller follicles showed lower rates ( 60%).

Lately new triggering protocols have emerged aiming to improve the proportion of mature oocytes at the time of retrieval. The aim of this study is to learn the effects of the dual triggering compared to the standard hCG triggering on the oocyte development and quality as a function of the follicle size

DETAILED DESCRIPTION:
Controlled ovarian hyperstimulation is critical to assisted reproduction because it increases the number of oocytes undergoing development. The medications, designed to override the selection of a single dominant follicle, drive multiple antral follicles into the growth phase. These follicles grow at different rates, and management is guided by their size rather than their competence. Human chorionic gonadotropin (hCG) is usually used as a surrogate LH surge to induce luteinization of the granulosa cells, final oocyte maturation and resumption of meiosis. This treatment is therefore based on an assumption that follicular size predicts the developmental competence of the oocyte. The outcome, is that only a portion of the oocytes will be competent for fertilization and development into viable embryos.

Studies have shown that the follicles greater in diameter was most likely to have a mature oocyte that was capable of fertilization and best suited for development into a high-quality embryo. Smaller follicles showed lower rates ( 60%).

Lately new triggering protocols have emerged aiming to improve the proportion of mature oocytes at the time of retrieval. Following the observations demonstrating comparable or even better oocyte\embryos quality following GnRHa, compared to hCG trigger, and the different effects of LH and hCG on the downstream signaling of the LH receptor, GnRHa is now offered concomitant to the standard hCG trigger dose to improve oocyte/embryo yield and quality. To the best of our knowledge, no studies have been done comparing the effect of the dual triggering on the amount of larger follicles per cycle and its effect on oocyte maturation.

The aim of this study is to learn the effects of the dual triggering compared to the standard hCG triggering on the oocyte development and quality as a function of the follicle size

Material and Methods A prospective cohort study including all women on antagonist protocol for controlled ovarian hyper stimulation with triggering using Ovitrelle ( hCG 250 mcg) or dual triggering - Ovitrelle ( Hcg 250 mcg) + Decapeptyl ( GnRH Agonist 0.1 mg*2 ).

As practiced at the IVF clinic, individuals will be monitored with transvaginal ultrasound and blood samples for hormonal profile ( including Estradiol, Progesteron, FSH). The decision to administer hCG or Dual triggering will be based on physician judgment, and the timing will be based on the lead follicular cohort, usually with at least two follicles measuring 18 mm for maximal diameter. A transvaginal, ultrasound-guided follicular aspiration will be conducted 36 hours after triggering administration. At retrieval, each follicle will be measured before aspiration. Follicles will be divided into five arbitrary follicular groups according to their maximal dimensional size: >18 mm, 16 to 18 mm, 13 to 15 mm, 10 to 12 mm, and <10 mm. Following identification, the follicles will be aspirated. Microscopic examination of the follicular aspirates will be performed by the embryologist. Once the oocytes will be identified, they will be collected and organized according to follicle size. Oocytes will be fertilized using conventional insemination or intracytoplasmic sperm injection (ICSI) . Each embryo will be cultured and evaluated after 72 hours.

Day-3 embryo grading, based on cellular cleavage and fragmentation, will be recorded separately. Fragmentation will be scored by the degree of fragmentation proportional to the whole embryo volume: 1, no fragmentation; 2, <10%; 3, 10% to 25%; 4, 25% to 50%; 5, >50%. The information for each oocyte, starting from the follicular size, will be followed through all laboratory procedures including insemination, oocyte stripping for ICSI, ICSI, pronuclear assessment, embryo culture, and embryo transfer.

Data will be collected from the medical file of each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age- 18-45
2. Antagonist protocol
3. Triggering: A- with Ovitrelle ( HCG) 250 mcg B- with dual triggering - Ovitrelle ( HCG) 250 mcg + Decapeptyl ( GnRH Agonist ) 0.1 mg*2

Exclusion Criteria:

1. Endometriosis
2. Known mutation of Fragile X

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women during IVF treatment
Enrollment: 200 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Oocyte retrieved in each of the follicular size groups | Through study completion, an average of 1 year
  Number of oocyte retrieved in each of the follicular groups divided according to the maximal dimensional size

SECONDARY OUTCOMES:
Metaphase II oocytes (MII) | Through study completion, an average of 1 year
  Oocyte undergone nuclear maturation -Metaphase II oocytes (MII)
Fertilization rate | Through study completion, an average of 1 year
  Fertilization rate ( 2 pronuclear)
Top Quality Embryo | Through study completion, an average of 1 year
  Top Quality Embryo - Day-3 embryo with 3-4 cells with of to 15% fragmentation rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing the data

REFERENCES:
- [Result] Miller KF, Goldberg JM, Falcone T. Follicle size and implantation of embryos from in vitro fertilization. Obstet Gynecol. 1996 Oct;88(4 Pt 1):583-6. doi: 10.1016/0029-7844(96)00241-4. PMID 8841223
- [Result] Orvieto R. Triggering final follicular maturation-hCG, GnRH-agonist or both, when and to whom? J Assist Reprod Genet. 2016 Oct;33(10):1415-1416. doi: 10.1007/s10815-016-0775-4. Epub 2016 Jul 22. No abstract available. PMID 27448022
- [Result] Andersen CY. Characteristics of human follicular fluid associated with successful conception after in vitro fertilization. J Clin Endocrinol Metab. 1993 Nov;77(5):1227-34. doi: 10.1210/jcem.77.5.7521343.
- [Result] Rosen MP, Shen S, Dobson AT, Rinaudo PF, McCulloch CE, Cedars MI. A quantitative assessment of follicle size on oocyte developmental competence. Fertil Steril. 2008 Sep;90(3):684-90. doi: 10.1016/j.fertnstert.2007.02.011. Epub 2008 Feb 4. PMID 18249377
- [Result] Bergh C, Broden H, Lundin K, Hamberger L. Comparison of fertilization, cleavage and pregnancy rates of oocytes from large and small follicles. Hum Reprod. 1998 Jul;13(7):1912-5. doi: 10.1093/humrep/13.7.1912. PMID 9740448